CLINICAL TRIAL: NCT03069287
Title: Feasibility and Acceptability of Integrating Family Caregiver Support Into Cancer Clinical Trials
Brief Title: Integrating Family Caregiver Support Into Cancer Clinical Trials
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding and resources
Sponsor: Saint John's Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: JWCI-17-0102
Record Dates: First submitted 2017-02-27; First posted 2017-03-03 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Cancer; Clinical Trials; Caregivers
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient-caregiver dyads (Experimental): Dyads will include family caregivers and patients with a diagnosis of cancer who agreed to participate in a therapeutic clinical trial.
  Interventions: Behavioral: Benjamin Rose Institute (BRI) Care Consultation™ Program

INTERVENTIONS:
Behavioral: Benjamin Rose Institute (BRI) Care Consultation™ Program — The BRI Care Consultation™ can be delivered via face-to-face contact, telephone, mail, and/or email by a Care Consultant and caregiver who assists with daily activities, tasks, and health-related issues. BRI CareConsultation™ uses a secure, web-based Care Consultation Information System (CCIS) to guide the delivery of the intervention.

SUMMARY:
The aim of this study is to assess the effects of integrating family caregiver support into cancer clinical trials on the well-being of the caregiver, the care-recipient and on the cancer clinical trial system.

DETAILED DESCRIPTION:
The aim of this study is to assess the effects of integrating family caregiver support into cancer clinical trials on the well-being of the caregiver, the care-recipient and on the cancer clinical trial system. This study will allow us to examine the benefit of adding a personalized support program for the family caregiver of a patients participating in a cancer clinical trial. Findings will assist in strengthening patient/caregiver-centered care management and support programs developed to enhance the quality of life of patients with cancer and the caregivers, reduce barriers to clinical recruitment, and improve retention in clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* dyad must be at least 18 years of age,
* patient is enrolled or expressed intent to enroll in a therapeutic cancer clinical trial
* caregiver is a self-identified primary caregiver,
* able to speak, read, and understand English,
* willing to participate in completion of surveys, and
* co-residence

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-07-10 (Actual); Primary Completion 2023-02-14 (Actual); Study Completion 2023-02-14 (Actual)

PRIMARY OUTCOMES:
Absolute change in the Caregiver Reaction Assessment (CRA) score | 1 year
  Caregiver Reaction Assessment (CRA) will be used to measure caregiver burden. The instrument was designed as a questionnaire with Likert-type responses ranging from strongly agree (1) to strongly disagree. The 24 items form 5 distinct unidimensional subscales that include: family burden (lack of family support; 5 items), financial burden (struggle with bills; 3 items), health burden (caregivers' health decline; 4 items), schedule burden (disruption of daily tasks; 5 items), and caregiving esteem (7 items), a positive subscale that measures enjoyment and importance of caregiving. A higher score on the caregiver's esteem subscale indicates a more positive effect of caregiving while higher scores on the other subscales indicate greater negative effects of caregiving in those domains
Absolute change in the scores for the assessment domains included in the Ben Rose Institute (BRI) care consultation program | 1 year
  Assessment of multiple caregiver and patient domains addressed by the BRI Care Consultation program

SECONDARY OUTCOMES:
Absolute change in the Functional Assessment of Cancer Therapy - General (FACT-G) score | 1 year
  Assesses patient quality of life. There are 27 questions, each of which is answered using a 5-point scale ranging from 0 (Not at all) to 4 (Very much). Questions are phrased so that higher numbers indicate a better health state.
Absolute change in Patient Reported Outcomes- Common Toxicity Criteria for Adverse Events (PRO-CTCAE) scores | 1 year
  The Patient Reported Outcome-Common Toxicity Criteria for Adverse Events (PRO-CTCAE) assesses patient quality of life. PRO-CTCAE items evaluate the symptom attributes of frequency, severity, interference, amount, presence/absence. Each symptomatic AE is assessed by 1-3 attributes. Responses for each attribute (frequency, severity, and/or interference of symptoms) are scored from 1 to 5 with 1+ mild and 5 = death.
  1. - Mild
  2. - Moderate
  3. - Severe
  4. - Life-threatening
  5. - Death

CONTACTS AND LOCATIONS:
Locations (1):
- John Wayne Cancer Institute at Providence Saint John's Health Center, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Saria MG, Courchesne N, Evangelista L, Carter J, MacManus DA, Gorman MK, Nyamathi AM, Phillips LR, Piccioni D, Kesari S, Maliski S. Cognitive dysfunction in patients with brain metastases: influences on caregiver resilience and coping. Support Care Cancer. 2017 Apr;25(4):1247-1256. doi: 10.1007/s00520-016-3517-3. Epub 2016 Dec 5. PMID 27921222
- [Background] Saria MG, Nyamathi A, Phillips LR, Stanton AL, Evangelista L, Kesari S, Maliski S. The Hidden Morbidity of Cancer: Burden in Caregivers of Patients with Brain Metastases. Nurs Clin North Am. 2017 Mar;52(1):159-178. doi: 10.1016/j.cnur.2016.10.002. PMID 28189161